CLINICAL TRIAL: NCT00339209
Title: Prospective Lung Transplant Database for Genetic Research
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905184; 05-E-N184
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-13

CONDITIONS: Lung Transplantation Rejection
Keywords: Genetic Polymorphisms; Acute Rejection; Bronchiolitis Obliterans Syndrome; Transplant Rejection; Innate Immunity; Lung Transplantation Rejection
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

SUMMARY:
This study will create a database of clinical and biological research for use in future studies, with information obtained from lung transplant recipients. The database will consist of genetic material and clinical outcomes to be used in future genotyping studies, that is, studies regarding the genetic makeup of individuals. Lung transplantation has become an important option for patients with advanced lung disease. More than 10,000 patients have received them to date, and about 1,200 transplant operations are performed worldwide each year. Although short-term survival has continued to improve, the 5-year survival rate is less than 50 percent. Most post transplant deaths are directly or directly caused by chronic lung rejection, a condition of scarring that worsens lung function.

Patients evaluated for lung transplants at Duke University Medical Center may be eligible for this study.

For developing the database, a small amount of blood, about 3 tablespoons, will be collected from patients. Blood collection for the research will be done at the same time as blood is drawn for necessary tests. The blood cells and DNA (which contains genetic material) will be isolated for analysis. Patients' DNA samples collected will be identified by a code, and all other identifying information will be removed. Patients may be asked to donate additional blood samples after their lung transplant if researchers would like to reexamine their blood.

This study will not have a direct benefit for participants. However, during the study, if it is found that any patients have an inherited risk for a disease likely to cause early death if the disease is not treated, then the researchers will attempt to notify those patients. Overall, it is hoped that information gained during this study will help medical professionals to learn more about immune activation and to see how the reactivity of lung transplant patients changes over time. If specific genetic risks could be identified, it might lead to individualized treatments that work on the immune system. Short-term and long-term survival of lung transplant recipients may thus be improved.

DETAILED DESCRIPTION:
Lung transplantation has emerged as a viable therapeutic option in the care of patients with advanced pulmonary parenchymal and pulmonary vascular disease. Currently, over 10,000 patients have received lung transplantation with approximately 1200 transplant operations performed worldwide each year. Short-term survival after lung transplantation has continued to improve since the widespread application of this procedure and one-year survival at most centers now approaches 80%. Unfortunately, long-term outcomes after lung transplantation are disappointing with five-year survival below 50%. Most posttransplant deaths are due directly or indirectly to the development of acute or chronic rejection. Acute rejection is defined by the presence of perivascular mononuclear inflammatory cells. Obliterative bronchiolitis (OB) describes fibrosis and obliteration of the small to medium size bronchioles, the histological manifestation of chronic lung rejection. Bronchiolitis obliterans syndrome (BOS) is thought to correlate with the development of histological OB when other causes of allograft dysfunction have been excluded. The diagnosis of OB is based primarily on a decline in spirometry with exclusion of alternative diagnoses with bronchoscopy and biopsy, i.e. development of clinical BOS. Since the introduction of BOS nomenclature, numerous studies have validated the clinical and prognostic importance of this syndrome and verified its correlation with histological OB.

Chronic rejection describes a histological pattern of fibrous obliteration of endothelial or epithelial structures in the allograft. A similar pattern of histological fibrosis is observed in all types of solid organ transplants (e.g., obliterative arteriopathy in heart transplant, BOS in lung transplant), and occurs despite the use of currently available, primarily T-cell based, immune suppression. The rates of chronic rejection vary considerably with the type of organ transplanted. By five years after transplantation histological fibrosis occurs in approximately 20% of kidney, 40% of heart and 60-80% of lung recipients. Thus, lung transplantation is characterized by an unusually high incidence of chronic graft rejection manifest as BOS.

Because of the high rate of acute and chronic lung transplant rejection, research designed to better correlate clinical outcomes with the genetic risks for rejection is critical to improving patient outcomes. We recently completed a study that demonstrated two single nucleotide polymorphisms (SNPs) Asp299Gly and Thr399Ile (polymorphisms of the human Toll 4 gene associated with endotoxin hyporesponsiveness) were associated with decreased acute rejection after lung transplantation.

We hypothesize that other SNPs associated with either increased or decreased innate or adaptive immune activation will be critical to determining the clinical outcome with regards to acute and chronic rejection after lung transplant. If specific genetic risks for rejection after transplant could be identified, this might lead to highly tailored immunosuppressive regimens and improved clinical outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients evaluated for lung transplant at Duke University Medical Center will be eligible for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-06-23; Study Completion 2007-04-13

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina

REFERENCES:
- [Background] Tazelaar HD, Yousem SA. The pathology of combined heart-lung transplantation: an autopsy study. Hum Pathol. 1988 Dec;19(12):1403-16. doi: 10.1016/s0046-8177(88)80233-8. PMID 3142814